CLINICAL TRIAL: NCT05714228
Title: Validation of the EuroSCORE II in Open and Trans-catheter Mitral Valve Repair.
Status: Completed | Type: Observational
Sponsor: Michele De Bonis (Other)
Responsible Party: Sponsor-Investigator, Michele De Bonis, Chief of Cardiac Surgery of Advanced and Research Therapies, Ospedale San Raffaele
Organization: Ospedale San Raffaele (Other)
Other Study IDs: VEOT-MVR
Record Dates: First submitted 2023-01-27; First posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Mitral Valve Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgical repair
  Interventions: Procedure: Surgical Mitral Valve Repair
- Transcatheter repair
  Interventions: Procedure: Transcatheter Mitral Valve Repair

INTERVENTIONS:
Procedure: Surgical Mitral Valve Repair — Mitral valve is repaired using open surgical approach
  Groups: Surgical repair
Procedure: Transcatheter Mitral Valve Repair — Mitral valve is repaired using Mitraclip transcatheter device
  Groups: Transcatheter repair

SUMMARY:
The EuroSCORE II is widely used to predict 30-day mortality in patients undergoing open and trans-catheter cardiac surgery

* However, it has not been validated in patients undergoing surgical or trans- catheter mitral valve repair.
* The aim of this study is to evaluate the predictive value of the EuroSCORE II in estimating 30-day mortality in a large cohort of patients undergoing surgical and trans-catheter repair by means of Mitraclip implantation.

Methods

* Institutional database retrospective review for surgical mitral repair and MitraClip implantation.
* Time frame: January 2012-December 2019
* 2793 patients identified; Euroscore II 1.3% [0.6%-2%]
* Survival after hospital discharge was assessed by outpatients visit, usually done 2 months after the index procedure.

Statistical analysis

* Receiver operating characteristic (ROC) curves were used to determine the cut-offs of Euroscore II. ROC Area Under the Curve (AUC) values varies between 0 and 1, where 0.5 denotes a bad diagnostic test and 1 denotes an excellent diagnostic test.
* The maximum Youden's Index (J=sensitivity + specificity - 1) was employed to define the optimal cut-point.
* ROC curves were repeated for surgical and MitraClip patients separately, and for primary and secondary etiology as well.

ELIGIBILITY:
Inclusion Criteria:

* Patients undewent mitral valve repair with an open surgical approach, also in association with concomitant procedures (for example, but not limited to, aortic valve replacement, tricuspid repair, etc.)
* Patients undergoing transcatheter mitral valve repair with MitraClip implantation
* Patients operated on at the U.O. of Cardiac Surgery at the San Raffaele Hospital from January 2012 to December 2019

Exclusion Criteria:

* Patients underwent mitral valve replacement with prosthesis
* Cardiac surgery patients not eligible for mitral valve surgery
* Patients undergoing mitral implantation, both open and transcatheter, of devices in experimental clinical study (e.g., but not limited to, adjustable rings and neocords, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent surgical or transcatheter mitral valve repair
Sampling Method: Non-Probability Sample
Enrollment: 2645 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
Euroscore II overall predictive power | 30 days postop
Euroscore II predictive power for surgery | 30 days postop
Euroscore II predictive power for transcatheter | 30 days postop

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No